CLINICAL TRIAL: NCT04476082
Title: Analysis of Nutritional Status in Patients With Malignant Tumor Diseases of the Gastrointestinal Tract
Brief Title: Nutrition in Gastrointestinal Tumors
Acronym: NutriGIT
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 071/20
Record Dates: First submitted 2020-06-29; First posted 2020-07-17 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Oesophageal Cancer; Colon Cancer; Liver Cancer; Rectal Cancer; Bile Duct Cancer; GIST, Malignant; Neuroendocrine Tumors; Small Intestine Cancer; Gastric Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Liver Neoplasms; Rectal Neoplasms; Bile Duct Neoplasms; Gastrointestinal Stromal Tumors; Neuroendocrine Tumors; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Plasma, Faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initial Diagnosis: Patients with initial diagnosis of a malignant condition of the gastrointestinal tract planned to receive cytostatic treatment.
  Interventions: Other: No intervention - observational study only
- Ongoing Cytostatic Treatment: Patients with a malignant condition of the gastrointestinal tract already receiving cytostatic treatment.
  Interventions: Other: No intervention - observational study only

INTERVENTIONS:
Other: No intervention - observational study only — No intervention - observational study only

SUMMARY:
Malnutrition and loss of muscle mass frequently occur in patients undergoing chemotherapy and can negatively effect therapy outcome. Especially patients with cancer of the gastrointestinal tract are often affected by malnutrition. Therefore, this study aims to examine changes in nutritional status of patients with cancer of the gastrointestinal tract during chemotherapy. Findings of this study will help to improve nutritional treatment of patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Malnutrition and sarcopenia are common complications in patients with malignant diseases of the gastrointestinal tract. During chemotherapy there is a high risk of further impairment of nutritional status due to anorexia, nausea, emesis and other gastrointestinal conditions that adversely impact food assimilation or absorption. Findings on changes of nutritional status during chemotherapy are scarce but of paramount importance for adequate nutrition therapy. Therefore, this study aims to provide a detailed description of changes in nutritional status of patients with a malignant condition of the gastrointestinal tract during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis of a malignant condition of the gastrointestinal tract planned to receive cytostatic treatment.
* ongoing cytostatic treatment of a known malignant condition of the gastrointestinal tract

Exclusion Criteria:

* pregnancy
* history of any other malignant tumor disease
* inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at University Medicine Greifswald (Northeast Germany). Patients with initial diagnosis of a malignant condition of the gastrointestinal tract planned to receive cytostatic treatment will be identified in the gastrointestinal ward of the hosptial. Recruitment of patients receiving cytostatic treatment of a known malignant condition of the gastrointestinal tract will take place in the hospital's cancer day unit.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of Malnutrition According to the Global Leadership Initiative on Malnutrition criteria (GLIM criteria) | 3 months after study enrollment
  Change in prevalence of malnutrition according to the GLIM criteria

SECONDARY OUTCOMES:
Prevalence of Malnutrition According to the European Society for Clinical Nutrition and Metabolism criteria (ESPEN criteria) | 3 months after study enrollment
  Change in prevalence of malnutrition according to the ESPEN criteria
Skeletal Muscle Mass | 3 months after study enrollment
  Changes in the skeletal muscle mass measured by Bioelectrical Impedance Analysis (BIA)
Fat Free Mass | 3 months after study enrollment
  Changes in the fat free mass measured by Bioelectrical Impedance Analysis (BIA)
Fat Mass | 3 months after study enrollment
  Changes in the fat mass measured by Bioelectrical Impedance Analysis (BIA)
Total Body Water | 3 months after study enrollment
  Changes in the total Body water measured by Bioelectrical Impedance Analysis (BIA)
Extracellular Water | 3 months after study enrollment
  Changes in the total extracellular water measured by Bioelectrical Impedance Analysis (BIA)
Phase Angle | 3 months after study enrollment
  Changes in the phase angle measured by Bioelectrical Impedance Analysis (BIA)
Body Weight | 3 months after study enrollment
  Changes in body weight measured in kilograms
Height | 3 months after study enrollment
  Changes in height measured in meters
Body Mass Index | 3 months after study enrollment
  Changes in body mass index in kg/m^2 (calculated from the values obtained for body weight and height)
Waist Circumference | 3 months after study enrollment
  Changes in waist circumference measured in centimeters
Hip Circumference | 3 months after study enrollment
  Changes in hip circumference measured in centimeters
Waist-to-Hip Ratio | 3 months after study enrollment
  Changes in waist-to-hip ratio (calculated from the values obtained for waist and hip circumference)
Upper Arm Circumference | 3 months after study enrollment
  Changes in upper arm circumference measured in centimeters
Triceps Skinfold Thickness | 3 months after study enrollment
  Changes in triceps skinfold thickness measured in millimeters
Muscle Strength | 3 months after study enrollment
  Changes in muscle strength measured by a handgrip strength dynamometer
Muscle Function | 3 months after study enrollment
  Changes in muscle function measured by a 4-m gait speed test
Sarcopenia According to the European Working Group on Sarcopenia in Older People 2 criteria (EWGSOP2 criteria) | 3 months after study enrollment
  Change in prevalence of sarcopenia according to the EWGSOP2 criteria
Energy Intake | 3 months after study enrollment
  Changes in energy intake assessed by 3-day weighed dietary record
Protein Intake | 3 months after study enrollment
  Changes in protein intake (in g/day) assessed by 3-day weighed dietary record
Carbohydrate Intake | 3 months after study enrollment
  Changes in carbohydrate intake (in g/day) assessed by 3-day weighed dietary record
Fat Intake | 3 months after study enrollment
  Changes in fat intake (in g/day) assessed by 3-day weighed dietary record
Dietary Fiber Intake | 3 months after study enrollment
  Changes in dietary fiber intake (in g/day) assessed by 3-day weighed dietary record
Physical Activity | 3 months after study enrollment
  Changes in metabolic equivalent of task per day and activity level are assessed by employment of the German version of the International Physical Activity Questionnaire (IPAQ) Short Form
Complete Blood Count | 3 months after study enrollment
  Changes in complete blood count
Albumin | 3 months after study enrollment
  Changes in plasma concentration of albumin
Aspartate Transaminase | 3 months after study enrollment
  Changes in plasma concentration of aspartate transferase
Alanine Aminotransferase | 3 months after study enrollment
  Changes in plasma concentration of alanine aminotransferase
Gamma-glutamyl Transferase | 3 months after study enrollment
  Changes in plasma concentration of gamma-glutamyl transferase
Bilirubin | 3 months after study enrollment
  Changes in plasma concentration of bilirubin
Creatinine | 3 months after study enrollment
  Changes in plasma concentration of creatinine
Urea | 3 months after study enrollment
  Changes in plasma concentration of urea
C-reactive Protein | 3 months after study enrollment
  Changes in plasma concentration of C-reactive protein
Plasma Metabolome | 3 months after study enrollment
  Changes in plasma metabolome
Plasma Transcriptome | 3 months after study enrollment
  Changes in plasma transcriptome
Intestinal Microbiome | 3 months after study enrollment
  Changes in intestinal microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Aghdassi, Professor, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany